CLINICAL TRIAL: NCT01486381
Title: A Multi-national, Multi-centre, Open-labelled Extension Study Assessing the Long-term Safety of Biphasic Insulin Aspart 30 (BIAsp 30) in Young Diabetic Subjects With Type 1 Diabetes Mellitus Previously Treated in BIAsp-1240
Brief Title: Long Term Safety of Biphasic Insulin Aspart 30 in Juveniles With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1459
Record Dates: First submitted 2011-11-22; First posted 2011-12-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in South Africa. The aim of this trial is to investigate Long term safety of biphasic insulin aspart 30 in juveniles with type 1 diabetes previously treated in trial BIAsp-1240.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities according to local requirements. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* The subject must have completed the trial BIAsp-1240

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2002-03-20 (Actual); Primary Completion 2003-05-30 (Actual); Study Completion 2003-05-30 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycaemic episodes
Occurence of adverse events
Standard safety parameters: Haematology, biochemistry and vital signs

SECONDARY OUTCOMES:
HbA1c (glycosylated haemoglobin)
Blood glucose level at each time-point in the 8-point glucose profile
BMI (Body Mass Index)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- South Africa (2):
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com